CLINICAL TRIAL: NCT07223983
Title: Semaglutide Treatment for Alcohol Use Disorder After Metabolic and Bariatric Surgery: A Pilot Randomized Controlled Trial
Brief Title: Semaglutide (SEMA) for Alcohol Use Disorder (AUD) After Metabolic and Bariatric Surgery (MBS)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000039710
Record Dates: First submitted 2025-10-30; First posted 2025-11-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Alcohol Use Disorder; Weight Loss; Bariatric Surgery Patients
MeSH Terms: conditions — Alcoholism; Weight Loss | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to a medication (Semaglutide) or a wait-list control for three months with a subsequent six-month follow-up (total 9 months).
Who Masked: Outcomes Assessor
Masking Description: Post-treatment and six-month follow-up assessments will be completed by a study clinician that is blind to treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Experimental): Participants randomized to Semaglutide will be initiated on a 0.25 mg dose (injection) once weekly for 4 weeks (first month) with an escalation to 0.5 mg for the second month, and 1.0 mg in the final month. Participants will be on Semaglutide for three months total.
  Interventions: Drug: Semaglutide 1.0 mg
- Wait-list control (No Intervention): Participants randomized to wait-list control will be followed for three months but no treatment will be administered. At the conclusion of the study, participants in the wait list control group will be offered a three-month behavioral intervention to treat Alcohol Use Disorder, although this is not required.

INTERVENTIONS:
Drug: Semaglutide 1.0 mg — Participants randomized to Semaglutide will be initiated on a 0.25 mg dose (injection) once weekly for 4 weeks (first month) with an escalation to 0.5 mg for the second month, and 1.0 mg in the final month (three months total).
  Arms: Semaglutide

SUMMARY:
The purpose of this research study is to evaluate the feasibility of treating Alcohol Use Disorder with Semaglutide after metabolic and bariatric surgery in adults with overweight or obesity.

DETAILED DESCRIPTION:
This study aims to evaluate the feasibility and acceptability of treating Alcohol Use Disorder with Semaglutide after metabolic and bariatric surgery in adults with overweight/obesity. This study will also examine changes in alcohol use disorder and weight. It is hypothesized that the treatment will be feasible and acceptable to participants, and result in reductions in alcohol use and weight.

A recently published randomized controlled trial provided preliminary evidence that Semaglutide can reduce some alcohol craving and drinking outcomes; however, this has not been examined in individuals with a history of bariatric surgery who are at increased risk of alcohol misuse and Alcohol Use Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study (up to 9 months: 3-month treatment plus 6-month follow up)
* Age 18 and older
* Have a BMI ≥30 (or BMI ≥27 with a medical comorbidity) and BMI ≤50 kg/m2
* Have had laparoscopic Roux-en-Y gastric bypass or sleeve gastrectomy within the past three years
* Meet current DSM-5 criteria for Alcohol Use Disorder
* Be an otherwise healthy subject without uncontrolled medical problems, as determined by the study physician and medical co-investigators
* Read, comprehend, and write English at a sufficient level to complete study-related materials
* For females of reproductive potential: use of highly effective contraception and agreement to use such a method during study participation

Exclusion Criteria:

* Any of the following: myocardial infarction, stroke, hospitalization for unstable angina, or transient ischemic attack within the past 60 days prior to screening
* History or presence of chronic or recurrent pancreatitis
* History of malignant neoplasms within the past 5 years prior to screening
* Personal or family history of medullary thyroid carcinoma or in patients with Multiple Endocrine Neoplasia syndrome type 2
* Is currently using other medications for weight loss or other GLP-1 receptor agonists
* Has a history of allergy or sensitivity to Semaglutide
* Has a co-existing psychiatric condition that requires hospitalization or more intensive treatment (such as bipolar mood disorders, psychotic illnesses, or severe depression)
* Has untreated hypertension with a seated systolic blood pressure > 160 mmHg, diastolic blood pressure > 100 mmHg, or heart rate > 100 beats/minute
* Has current uncontrolled hypertension
* Has current uncontrolled Type I or Type II diabetes mellitus
* Has untreated hypothyroidism with a TSH > 1.5 times the upper limit of normal for the test laboratory with repeat value that also exceeds this limit
* Has active gallbladder disease
* Has a history of severe renal, hepatic, neurological, chronic pulmonary disease, or any other unstable medical disorder
* Has a recent history of substance use disorder (with the exception of cannabis or tobacco use disorder) within the past 12 months
* Is currently engaging in other treatment for Alcohol Use Disorder or making intentional efforts to quit alcohol use
* Is currently participating in another clinical study in which the subject is or will be exposed to an investigational or a non-investigational drug or device
* Is breast-feeding, pregnant, or not using a reliable form of birth control
* Reports active suicidal or homicidal ideation
* Any disorder, unwillingness or inability, not covered by any of the other exclusion criteria which, in the investigator's opinion, might have jeopardized the participant's safety or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Percent weight change | Baseline, Week 12, 6-month follow-up
  Percent weight change will be calculated. Negative values are indicative of weight loss. Positive values are indicative of weight gain.
Mean drinks per calendar day to assess alcohol use | Baseline, Week 4, Week 8, Week 12, 6-month follow-up
  Mean drinks per calendar day will be assessed through timeline follow back interviews
Mean drinks per drinking day to assess Alcohol use | Baseline, Week 4, Week 8, Week 12, 6-month follow-up
  Mean drinks per drinking day will be assessed through timeline follow back interviews
Mean number of heavy drinking days to assess Alcohol use | Baseline, Week 4, Week 8, Week 12, 6-month follow-up
  Mean number of heavy drinking days will be assessed through timeline follow back interviews
Mean number of drinking vs abstinent days to assess Alcohol use | Baseline, Week 4, Week 8, Week 12, 6-month follow-up
  Mean number of drinking vs abstinent days will be assessed through timeline follow back interviews

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Ivezaj, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hendershot CS, Bremmer MP, Paladino MB, Kostantinis G, Gilmore TA, Sullivan NR, Tow AC, Dermody SS, Prince MA, Jordan R, McKee SA, Fletcher PJ, Claus ED, Klein KR. Once-Weekly Semaglutide in Adults With Alcohol Use Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2025 Apr 1;82(4):395-405. doi: 10.1001/jamapsychiatry.2024.4789. PMID 39937469